CLINICAL TRIAL: NCT05694585
Title: Effect of Continuous Infusion of Esmolol on Perioperative Stress Reaction in Patients Undergoing Airway Intervention
Brief Title: Effect of Esmolol on Perioperative Stress Reaction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiumei Song (Other)
Responsible Party: Sponsor-Investigator, Xiumei Song, Associate chief physician, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YXLL-KY-2022(107)
Record Dates: First submitted 2023-01-05; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Esmolol; Stress Reaction; Airway Obstruction; Catecholamine; Overproduction
Keywords: continuous infusion
MeSH Terms: conditions — Fractures, Stress; Airway Obstruction | interventions — esmolol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- esmolol group (Experimental): esmolol group: esmolol 50 μg/kg /min were intravenously administered before Operation beginning. If HR（heart rate）is greater than 90 beats/min, esmolol 50μg/kg /min is added each time, with interval more than 5 min and the peak value is 200 μg/kg/min. If the heart rate is lower than 60 times/minute, Stop medication.
  Interventions: Drug: Esmolol
- Saline solution (Placebo Comparator): Saline group: saline 50 μg/kg /min were intravenously administered before Operation beginning. If HR（heart rate）is greater than 90 beats/min, saline 50μg/kg /min is added each time, with interval more than 5 min and the peak value is 200 μg/kg/min. If the heart rate is lower than 60 times/minute, Stop medication.
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Esmolol — Esmolol 50μg/kg /min is intravenously administered before Operation beginning. If HR（heart rate）is greater than 90 beats/min, esmolol 50μg/kg/min is added each time, with interval more than 5 min and the peak value is 200 μg/kg/min. If the heart rate is lower than 60 times/minute, Stop medication.
  Other Names: Esmolol hydrochloride
  Arms: esmolol group
Drug: saline — Saline 50μg/kg /min were iv administered before Operation beginning. If HR（heart rate）is greater than 90 beats/min, saline 50μg/kg/min is added each time, with interval more than 5 min and the peak value is 200 μg/kg/min. If the heart rate is lower than 60 times/minute, Stop medication.
  Other Names: 0.9% sodium chloride injection solution
  Arms: Saline solution

SUMMARY:
The goal of this clinical trial is to observe the effect of low dose continuous infusion of esmolol on perioperative stress response in patients undergoing airway intervention .

DETAILED DESCRIPTION:
Airway intervention is known to activate stress response and release catecholamines resulting in severe hemodynamic instability. Various techniques which are recommended to prevent the stress response include increasing the depth of anesthesia, improving surgical procedures and the use of various pharmacological agents. Esmolol blocks the action of the endogenous catecholamines, we plan low dose esmolol infusion decrease stress response and hemodynamic fluctuation during airway intervention.

46 patients scheduled airway intervention under general anesthesia were randomly divided into esmolol group and control group. esmolol 50μg/kg/min or saline 50μg/kg/min were iv administered before Operation beginning. If HR（heart rate）is greater than 90 beats/min, esmolol or saline 50μg/kg/min is added each time, with interval more than 5 min and the peak value is 200 μg/kg/min. If the heart rate is lower than 60 times/minute, Stop medication. Plasma level of Norepinephrine, epinephrine, and cortisol before induction of anesthesia and 30 minutes after beginning of operation were determined by high-performance liquid chromatography. Perioperative hemodynamics changes, extubation time, incidence of severe sinus bradycardia and bronchospasm were recorded.

ELIGIBILITY:
Inclusion criteria

1. American Society of Anesthesiologists (ASA) Physical Status I to III.;
2. Body mass index (BMI): 20-30 kg/m2;
3. Elective airway intervention under general anesthesia with jet ventilation，duration of operation less than 2hs;
4. Sign informed consent for clinical trial

Exclusion criteria

1. The patient and his or her family refused to participate in the study;
2. Severe respiratory or/cardiovascular or/ neurological disease, or/ hepatic or/renal dysfunction
3. Those who are allergic to the drugs used in this study;
4. Psychiatric history or with unstable mental state;
5. Patients with atrioventricular block
6. Patients with history of asthma
7. Patients now treated with β-adrenergic receptor blockers
8. Patients participating in other clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma norepinephrine levels | up to 30 minutes after beginning of operation
  level of Norepinephrine
Changes in plasma epinephrine levels | up to 30 minutes after beginning of operation
  level of epinephrine
Changes in plasma cortisol levels | up to 30 minutes after beginning of operation
  level of cortisol

SECONDARY OUTCOMES:
Hemodynamic changes ：Systolic blood pressure（SBP ） | from anesthesia induction to 30 minutes after remove the laryngeal mask
  Systolic blood pressure (SBP ) during perioperative period
Hemodynamic changes ：Diastolic blood pressure（ DBP） | from anesthesia induction to 30 minutes after remove the laryngeal mask
  Diastolic blood pressure（ DBP） during perioperative period
Hemodynamic changes ：Heart rate（HR） | from anesthesia induction to 30 minutes after remove the laryngeal mask
  Heart rate（HR） during perioperative period
Incidence of adverse reactions: Severe sinus bradycardia | from anesthesia induction to 30 minutes after remove the laryngeal mask
  Severe sinus bradycardia: HR<40 times/min during perioperative period
Incidence of adverse reactions: bronchospasm | from anesthesia induction to 30 minutes after remove the laryngeal mask
  Perioperative bronchospasm
Laryngeal mask airway (LMA) removal time | Duration from the end of anesthetics infusion to LMA removal
  Duration from the end of anesthetics infusion to LMA removal

CONTACTS AND LOCATIONS:
Overall Officials: Jinwan Guo, Master, Principal Investigator — Qianfoshan Hospital; Ling Dong, M.D., Principal Investigator — Qianfoshan Hospital; Yang Liu, M.D., Principal Investigator — Qianfoshan Hospital; Liang Guo, M.D., Principal Investigator — Qianfoshan Hospital

IPD SHARING:
Plan to Share IPD: Yes
demographic data，statistical data，study protocol
Supporting Information: Study Protocol, SAP
Time Frame: after 2024/1/1
Access Criteria: undecided

REFERENCES:
- [Background] Lakhe G, Pradhan S, Dhakal S. Hemodynamic Response to Laryngoscopy and Intubation Using McCoy Laryngoscope: A Descriptive Cross-sectional Study. JNMA J Nepal Med Assoc. 2021 Jul 1;59(238):554-557. doi: 10.31729/jnma.6752. PMID 34508397
- [Background] Hoshijima H, Maruyama K, Mihara T, Boku AS, Shiga T, Nagasaka H. Use of the GlideScope does not lower the hemodynamic response to tracheal intubation more than the Macintosh laryngoscope: a systematic review and meta-analysis. Medicine (Baltimore). 2020 Nov 25;99(48):e23345. doi: 10.1097/MD.0000000000023345. PMID 33235101
- [Background] Mendonca FT, Silva SLD, Nilton TM, Alves IRR. Effects of lidocaine and esmolol on hemodynamic response to tracheal intubation: a randomized clinical trial. Braz J Anesthesiol. 2022 Jan-Feb;72(1):95-102. doi: 10.1016/j.bjane.2021.01.014. Epub 2021 Sep 25. PMID 34582903
- [Background] Efe EM, Bilgin BA, Alanoglu Z, Akbaba M, Denker C. Comparison of bolus and continuous infusion of esmolol on hemodynamic response to laryngoscopy, endotracheal intubation and sternotomy in coronary artery bypass graft. Braz J Anesthesiol. 2014 Jul-Aug;64(4):247-52. doi: 10.1016/j.bjane.2013.07.003. Epub 2013 Oct 25. PMID 24998108
- [Background] Hasegawa D, Sato R, Prasitlumkum N, Nishida K, Takahashi K, Yatabe T, Nishida O. Effect of Ultrashort-Acting beta-Blockers on Mortality in Patients With Sepsis With Persistent Tachycardia Despite Initial Resuscitation: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Chest. 2021 Jun;159(6):2289-2300. doi: 10.1016/j.chest.2021.01.009. Epub 2021 Jan 9. PMID 33434497